CLINICAL TRIAL: NCT04935853
Title: Marqueurs Pronostiques et prédictifs de réponse Aux Traitements Chez Les Patients Atteints de Cancer Des Voies Biliaires : Cohorte Multicentrique ACABi PRONOBIL
Brief Title: Prognostic and Predictive Markers of Response to Treatment in Patients With Bile Duct Cancer: ACABi PRONOBIL Study
Status: Recruiting | Type: Observational
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Other Study IDs: ACABi PRONOBIL GB-115
Record Dates: First submitted 2021-05-28; First posted 2021-06-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Biliary Tract Cancer
Keywords: predictive; prognostic; biliary track cancer
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to identify prognosis and predictive markers of response to treatments (surgery, chemotherapy, targeted therapy,loco-regional treatments ) in patients with bile duct cancer. The effectiveness and tolerance of these treatments in current practice will also be evaluated.

DETAILED DESCRIPTION:
Bile duct cancers are a heterogeneous group of rare tumors with a poor prognosis. Surgery is the only curative modality for localized forms. Chemotherapy is the standard treatment in advanced forms. Identification of prognostic and predictive markers to better stratify patients and to guide therapeutic decisions is a major issue. It is retro-prospective (diagnosis between 2003 and 2021) and prospective (diagnosis between 2021 and 2030) multi-center, cohort study. Follow-up for 10 years from initial cancer diagnosis will be done.

Follow-up is retrospective only for patients operated on or diagnosed in the past for more than 10 years, and retro-prospective for operated patients or diagnosed in the past for less than 10 years.

The data collected for each patient are available during the life cycle of this clinical trial to fulfil an educational requirement (e.g. a doctoral thesis) upon request and authorization from the study committee and the study sponsor (GERCOR).

ELIGIBILITY:
Inclusion Criteria:

* All locations of primitives (intrahepatic CCA, extrahepatic CCA, adenocarcinoma of the gallbladder; ampullomas excluded)
* Age > 18 years
* Diagnosed between 2003 and 2030 (minimum follow-up 2 years)
* Written written non-opposition +/- signed informed consent for genetic studies (N.B.:

exemption requested for a deceased patient) N.B. Authorized inclusion in a therapeutic research protocol

Exclusion Criteria:

* Patient under guardianship, curatorship or legal protection
* Pregnant or breastfeeding women
* Any medical, psychological or social situation, which could prevent the compliance with the protocol according to the investigator's assessment
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retro-prospective (diagnosis between 2003 and 2020) and prospective (diagnosis between 2021 and 2030) cohorts of patients with Bile Duct Cancer
Sampling Method: Non-Probability Sample
Enrollment: 1350 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2030-06-01 (Estimated); Study Completion 2040-06-01 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with advanced bile duct cancer (BDC) experiencing overall survival (OS) less than 6 months | Up to 10 years from the date of initial cancer diagnosis (or until death if it occurs before 10 years)
  Identification of clinical and tumor predictive factors of overall survival (OS) (prognostic markers) in patients with advanced bile duct cancer (BDC).
  OS defined as a period between the start of treatment and death, whatever the cause.

SECONDARY OUTCOMES:
Rate of patients with localized bile duct cancer (BDC) experiencing overall survival (OS) less than 6 months | Up to 10 years from the date of initial cancer diagnosis (or until death if it occurs before 10 years)
  Identification of clinical and tumor predictive factors of overall survival (OS) (prognostic markers) in patients with bile localized BDC (operated).
  OS defined as a period between the start of treatment and death, whatever the cause.
Response rate | Up to 10 years from the date of initial cancer diagnosis (or until death if it occurs before 10 years)
  Assessment of treatments effects on the response rate (RECIST v 1.1, Choi).
Effect of treatments on secondary resection rate R0 of the primary tumor | From day of surgical intervention until 30 days
  Assessment of treatments on secondary resection rate R0 of the primary tumor
Effects of treatments on disease-free survival (DFS) | Up to 10 years; The months between surgery and the first documented recurrence, second cancer, or death from any cause
  Assessment of treatments effects on disease-free survival (DFS) in patients who underwent surgery.
Effects of treatments on progression-free survival (PFS) | Up to 10 years; The months between the start of treatment and the first progression or death, whatever be the cause
  Assessment of treatments effects on progression-free survival (PFS) in non-operated patients
Toxicities (Adverse events) experienced by patients | Up to 10 years from the date of initial cancer diagnosis (or until death if it occurs before 10 years)
  Evaluation of toxicity assessed by CTCAE v 5.0
The complications and postoperative mortality rates in patients who underwent surgery | From day of surgical intervention until 30 days; up to 10 years
  Assessment of the complications rate (Clavien classification) and of postoperative mortality in patients who underwent surgery

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Neuzillet, Dr, Principal Investigator — Institut Curie, Saint-Cloud
Locations (32):
- France (32):
  - CHU Hôpital Sud Amiens, Amiens
  - CHU Angers, Angers
  - CHU Besançon, Besançon
  - Hôpital Avicenne, Bobigny
  - CHU - Henri Mondor, Créteil
  - CHU Dijon, Dijon
  - CHU Grenoble, Grenoble
  - CHU Lille, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital Croix Rousse, Lyon
  - Hôpital Edouard Herriot, Lyon
  - Hôpital Privé Jean Mermoz, Lyon
  - Institut Paoli Calmette, Marseille
  - CHU Saint Eloi Montpellier, Montpellier
  - CHR Orléans, Orléans
  - Groupe Hospitalier Pitié Salpêtrière, Paris
  - Hôpital Ambroise Paré, Paris
  - Hôpital Cochin, Paris
  - Hôpital Saint Antoine, Paris
  - Hôpital Saint Louis, Paris
  - Institut Mutualiste Montsouris, Paris
  - Hôpital Haut Lévêque, Pessac
  - CHU Poitiers, Potiers
  - Hôpital Robert Debré -CHU Reims, Reims
  - Centre Eugène Marquis, Rennes
  - CHU Rouen Charles Nicolle, Rouen
  - Institut Curie, Saint-Cloud
  - CHU Saint Etienne, Saint-Etienne
  - CHU Rangueil, Toulouse
  - CHU Tours, Tours
  - CHRU Nancy Site Brabois, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Adamus N, Edeline J, Henriques J, Fares N, Lecomte T, Turpin A, Vernerey D, Vincens M, Chanez B, Tougeron D, Tournigand C, Assenat E, Delaye M, Manfredi S, Bouche O, Williet N, Vienot A, Blaise L, Mas L, Neuzillet C, Boileve A, Roth GS. First-line chemotherapy with selective internal radiation therapy for intrahepatic cholangiocarcinoma: The French ACABi GERCOR PRONOBIL cohort. JHEP Rep. 2024 Nov 20;7(2):101279. doi: 10.1016/j.jhepr.2024.101279. eCollection 2025 Feb. PMID 39897613